CLINICAL TRIAL: NCT00006825
Title: A Safety Study Of Doxil And Herceptin In Patients With Advanced Her-2 Overexpressing Breast Cancer
Brief Title: Liposomal Doxorubicin and Trastuzumab in Treating Women With Advanced Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068331; P30CA016087 (NIH); NYU-0012; ALZA-00-001-ii; NCI-G00-1878
Record Dates: First submitted 2000-12-06; First posted 2003-01-27 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

INTERVENTIONS:
Biological: trastuzumab
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining chemotherapy with monoclonal antibody therapy may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of liposomal doxorubicin and trastuzumab in treating women who have advanced breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity, including cardiac toxicity, of doxorubicin HCl liposome and trastuzumab (Herceptin) in women with advanced HER-2/neu-overexpressing breast cancer.
* Determine the efficacy of this regimen in these patients.

OUTLINE: Patients receive doxorubicin HCl liposome IV over 1 hour on day 1, followed by trastuzumab (Herceptin) IV over 30-90 minutes on days 1, 8, and 15. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven breast cancer

  * Metastatic disease OR
  * Locoregional relapse following optimal adjuvant therapy and regional treatment
  * HER-2/neu overexpression (3+ by immunohistochemistry OR gene amplification by FISH)
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 10 g/dL

Hepatic:

* SGOT and SGPT no greater than 3 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2 times ULN unless documented to be arising from bone
* Bilirubin no greater than 1.5 times ULN

Renal:

* BUN less than 1.5 times ULN
* Creatinine less than 1.5 times ULN

Cardiovascular:

* LVEF normal by radioisotope method
* No history of congestive cardiac failure, myocardial infarction, cardiac arrhythmia, or ischemic heart disease requiring medication

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No known sensitivity to benzyl alcohol
* No other prior malignancy except adequately treated nonmelanomatous skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Biologic therapy:

* Not specified

Chemotherapy:

* No prior doxorubicin greater than 240 mg/m2

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior radiotherapy to left breast or chest wall allowed

Surgery:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-07; Primary Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D. Volm, MD, Study Chair — NYU Langone Health
Locations (1):
- NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York, United States